CLINICAL TRIAL: NCT05196321
Title: Effects of Treatment With ENF (Electro Neuro Feedback) in the Reduction of Post-surgical Hematoma in Patients Undergoing Hip Replacement: Evaluation With Ultrasound Method
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: ENF PTA
Record Dates: First submitted 2021-11-25; First posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2021-11

CONDITIONS: Post-surgical Hematoma, Hip Replacement , Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: sessions with ENF (Electro Neuro Feedback). — The study evaluates patients with clinical evidence of post-surgical hematoma / seroma after hip replacement surgery. These patients will undergo ultrasound evaluation in the 4th (+/- 2) day post surgery, in which triaxial parameters of the hematoma will be measured. This evaluation will then be repeated after 5 treatment sessions with ENF (Electro Neuro Feedback).

SUMMARY:
The study evaluates patients with clinical evidence of post-surgical hematoma / seroma after hip replacement surgery. These patients will undergo ultrasound evaluation in the 4th (+/- 2) day post surgery, in which triaxial parameters of the hematoma will be measured. This evaluation will then be repeated after 5 treatment sessions with ENF (Electro Neuro Feedback). The patient will then be subjected to evaluation scales that allow to evaluate the subjective improvement of the state of well-being after treatment ENF (Electro Neuro Feedback) generates waveforms that change automatically when the impedance of the skin changes according to a compensation algorithm, i.e. according to Feedback (Feedback). T

ELIGIBILITY:
Inclusion Criteria:

* Gender: male and female
* Age: 35-85 years include
* Entry into the hospital rehabilitation program lasting at least 5 days following hip replacement surgery
* Absence in history of neurological or psychiatric disorders.
* Signature of the Informed Consent and consent to collaborate in all the procedures of the study

Exclusion Criteria:

* Presence of severe neurological / psychiatric pathologies
* to sign the Informed Consense
* of serious cardiological pathologies that can compromise patient safety
* of Pace Maker or spinal cord stimulators or other subcutaneous electronic instruments
* of active tumors in the treatment area

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population is made up of patients who have undergone hip prosthesis surgery with the presence of post-surgical hematoma who are included in the hospital rehabilitation program lasting at least 5 days following this intervention.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2023-07-20 (Estimated)

PRIMARY OUTCOMES:
change of post-surgical hematoma measured by ultrasound method with triaxial measurement after 5 treatment sessions with ENF | at the end of Cycle 5 ( every cycle during 5 days)

CONTACTS AND LOCATIONS:
Overall Officials: cristina beretta, Principal Investigator — IRCCS istituto ortopedico galeazzi -sede san siro
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi -San Siro, Milan, Italy